CLINICAL TRIAL: NCT02919774
Title: Biomarker Assessment of Pomaglumetad on Glutamate Targets: Proof of Clinical Mechanism of Action (POCM)
Brief Title: Pomaglumetad Effects on Glutamate Biomarkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marlene Carlson, Study Manager, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7285; 271201200007I-4-27100003-2 (NIH)
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Healthy Controls
MeSH Terms: interventions — poly(n-octyl methacrylate); pomaglumetad methionil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- POMA 40 mg BID (Experimental): 40 mg BID for 10 days
  Interventions: Drug: POMA
- POMA 160 mg BID (Experimental): 160 mg BID for 10 days
  Interventions: Drug: POMA
- Placebo (Placebo Comparator): Placebo BID for 10 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: POMA — Pomaglumetad ("POMA") is a mGluR 2/3 partial agonist
  Other Names: Pomaglumetad
  Arms: POMA 160 mg BID; POMA 40 mg BID
Drug: placebo — matching placebo tablets
  Other Names: placebo comparator
  Arms: Placebo

SUMMARY:
The study will evaluate the effects of the mGluR2/3 partial agonist LY2140023 (Pomaglumetad Methionil, "POMA") at selected doses on ketamine-stimulated glutamate release in prefrontal cortex as measured by pharmacoBOLD fMRI (also termed resting BOLD fMRI).

DETAILED DESCRIPTION:
This study evaluates the effects of POMA at selected doses on ketamine-stimulated glutamate increase in the prefrontal cortex hypothesized to simulate the synaptic dysregulation that occurs endogenously in the pathogenesis of schizophrenia. The purpose of this is: 1) to determine whether the low dose (40 mg BID) utilized in recent (failed) clinical trials is sufficient to engage the primary target and 2) whether a higher (160 mg BID) dose, representing the maximum tolerated dose of POMA, engages the target to a greater degree. This study will further validate pharmacoBOLD as biomarker of mGluR2/3 target engagement, permitting its future use in other glutamatergic drug development.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Capable of understanding the study procedures and able to provide informed consent
* Men and women must agree to use a reliable method of birth control during the study. Women who are post-menopausal or otherwise not of childbearing potential are also eligible

Exclusion Criteria:

* Current or past Axis I psychiatric history
* Positive urine toxicology
* History of recreational ketamine use, recreational PCP use, or an adverse reaction to ketamine. Subjects who have participated in prior research ketamine studies will be eligible. Subjects can have infusions not more frequently than biweekly, and not more than 1/month on average, therefore subjects entering the study will need to wait one month if they had a single infusion and 6 weeks if they have had two closely spaced infusions.
* History of first-degree relative with schizophrenia
* History of violence
* Presence or positive history of significant medical illness
* Presence or positive history neurological illness or any other disease/procedure/accident/intervention association with significant injury to or malfunction of the central nervous system (CNS) or history of significant head injury
* Pregnancy or breast feeding
* Metal implants, pacemaker, other metal or paramagnetic objects contained within the body
* Medicinal patch, unless removed prior to MRI scan
* Currently taking any psychotropic medication, including antidepressant medications, benzodiazepines, antipsychotic medications, mood stabilizers, anti-epileptic medications and stimulants.
* Claustrophobia
* Suicidal ideation with intent or plan in the 6 months prior to screening
* Weight > 86.95 kg (191.2 lbs)
* Subthreshold pharmacoBOLD response during screening ketamine infusion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
PharmacoBOLD change | Day 1 to Day 10
  pharmacoBOLD change, as summarized by the Amplitude measure

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | Day 1 to Day 10
  Clinical rating scale assessing common psychiatric symptoms
Clinician Administered Dissociative States Scale (CADSS) | Day 1 to Day 10
  Rates dissociative symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, MD, Principal Investigator — New York State Psychiatric Institute
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - New York University, New York, New York
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Submit to NDCT